CLINICAL TRIAL: NCT00069433
Title: Skills Training for Schizophrenia: Enhancing Outcomes
Brief Title: Enhancing the Outcome of Skills Training for People With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #4339; R01MH066362 (NIH); DSIR AT-SP
Record Dates: First submitted 2003-09-24; First posted 2003-10-09 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: Schizophrenia
Keywords: Psychotic Disorders
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Social skills and symptom management training

SUMMARY:
This study will determine the effectiveness of skills training in people with schizophrenia and the applicability of the acquired skills in the "real world."

DETAILED DESCRIPTION:
People with schizophrenia have a large number of social and symptom management training programs available to them. Studies suggest that these training programs are effective, but their generalizability and effectiveness in outpatient settings has not been thoroughly examined. This study will examine the treatment outcomes of a skills training approach in schizophrenic individuals taking antipsychotic medication.

Participants taking stable doses of risperidone, olanzapine, or quetiapine will be randomly assigned to receive either intensive symptom management and social skills training or group therapy for 12 months. A verbal memory test will be used to stratify the randomization procedure and to control for neurocognitive functioning.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder for > 5 years
* Use of stable dose risperidone, olanzapine, or quetiapine for at least 1 month with no planned medication changes
* Social Behavior Scale (SBS) score > 45
* Willing and able to provide informed consent

Exclusion Criteria:

* Intelligence Quotient < 70
* Use of more than one antipsychotic medication
* Use of benzodiazepines, tricyclic antidepressants, or anticholinergic medication commonly used to treat extrapyramidal symptoms
* Diagnostic and Statistical Manual (DSM)-IV criteria for alcohol or other substance dependence
* History of any traumatic brain injury leading to loss of consciousness for > 30 minutes
* Diagnosis of a comorbid medical condition that could interfere with antipsychotic medication treatment or the ability to complete the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60
Dates: Start 2001-04; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Hall-Brooke-The Center, Bridgeport, Connecticut
  - Hall-Brooke Behavioral Health Services, Westport, Connecticut